CLINICAL TRIAL: NCT03354078
Title: The Effect of Subcutaneous Tissue Closure Technique in Cesarean Section on Reducing Postoperative Wound Complications
Brief Title: Effect of Subcutaneous Tissue Closure on Wound Complications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aljazeera Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Cesarean section / sutures
Record Dates: First submitted 2017-11-19; First posted 2017-11-27 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Cesarean Section
Keywords: Cesarean section; Wound infection; Gapping
MeSH Terms: conditions — Wound Infection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interrupted sutures group (Active Comparator): This group in which closure of the subcutaneous layer is closed by interrupted sutures
  Interventions: Procedure: interrupted sutures; Procedure: continous sutures
- Continous sutures group (Active Comparator): subcutanous tissue layer is closed by continous sutures in this group
  Interventions: Procedure: interrupted sutures; Procedure: continous sutures

INTERVENTIONS:
Procedure: interrupted sutures — The way of closing subcutaneous tissue either by interrupted
Procedure: continous sutures — The way of closure of subcutanous tissue is by continous sutures

SUMMARY:
Only a small number of research studies evaluated the impact of various subcutaneous tissue and skin closure methods at cesarean section. In a meta-analysis a major decline in incision site rupture was revealed when suturing the subcutaneous tissue in women with a subcutaneous depth >2 cm.

DETAILED DESCRIPTION:
Postoperative wound complications are one of the great issues in cesarean section (CS) with an incidence ranging from 3% to 30%.1 Obesity, operative time, diabetes, age of the patient, anemia, associated infection (e.g chorioamnionitis), the use of internal monitoring, delayed labor with many vaginal examinations and reduced nutrition are recognized risk factors for wound infections.

Evaluating the various techniques for closure of the subcutaneous layer.

ELIGIBILITY:
Inclusion Criteria:

* All patients included in this research BMI ≥ 30, First cesarean section performed, no medical disorders with pregnancy e.g DM, HTN. All patients were subjected to full history taking, examination.

depth of subcutaneous tissue estimated by a special device used (sterilized operative ruler). number of sutures estimation

Exclusion Criteria:

* The following patients were excluded BMI <30, Previous CS, DM with pregnancy, HTN with pregnancy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant females
Enrollment: 400 (Actual)
Dates: Start 2017-06-18 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-23 (Actual)

PRIMARY OUTCOMES:
The number of participants who passed without postoperative complications | one month post cesarean section
  Describes how many participant willnot complain from wound seroma , wound erythema and wound infection

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Alalfy, M.s.c, Study Chair — Algazeerah hospital -Location (Giza -Egypt )
Locations (1):
- Algazeerah, Giza, Egypt

REFERENCES:
- [Derived] Alalfy M, Elgazzar A, Fares T, Nagy O, Ellithy A, Lasheen Y, Kamel A, Soliman M, Hassan A, Samy A, Taher AM, Ogila AI, Saad H, Salah H, Ramadan M, Nabil M, Hatem DL, Fikry M. Effect of subcutaneous tissue closure technique in cesarean section on postoperative wound complications in obese Egyptian women. J Matern Fetal Neonatal Med. 2019 Aug;32(15):2452-2459. doi: 10.1080/14767058.2018.1438399. Epub 2018 Feb 20. PMID 29415592